CLINICAL TRIAL: NCT04854564
Title: Identifying Perceived Barriers and Facilitators to Inform the Development of a Liver Transplantation Prehabilitation Intervention
Brief Title: Identifying Perceived Barriers and Facilitators Toward a Liver Transplantation Prehabilitation
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Haiyan Qu, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300007058
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Liver Transplant; Complications
Keywords: end-stage liver disease (ESLD); frailty; prehabilitation
MeSH Terms: conditions — End Stage Liver Disease; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- End-stage liver disease (ESLD) patients: These potential liver transplant candidates are patients with end-stage liver disease (ESLD) who have been assigned to the liver transplant waitlist.
  Interventions: Behavioral: Prehabilitation intervention
- Caregivers of potential liver transplant candidates: They are the primary caregivers for the patients.
  Interventions: Behavioral: Caregiver intervention

INTERVENTIONS:
Behavioral: Prehabilitation intervention — The investigators will identify participants' perceived important information to develop a prehabilitation intervention in this study. Prehabilitation intervention consisting of physical activities, nutrition, and stress management.
  Groups: End-stage liver disease (ESLD) patients
Behavioral: Caregiver intervention — The investigators will provide caregivers with variety of educational resources for patients experiencing ESLD.
  Groups: Caregivers of potential liver transplant candidates

SUMMARY:
The purpose of this study is to formally identify patient and caregiver perceived needs, barriers, and facilitators to inform the development of a home-based multimodal prehabilitation program for potential LT candidates.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants (patients and caregivers) giving written informed consent will be invited to participate in one of three research activities: interviews (n=10), nominal group technique meetings (n=64), or card-sorting and rating survey (n=40).

ELIGIBILITY:
Inclusion Criteria:

Liver transplant (LT) candidates are:

* Adult ESLD patients (age=19-74 years) who are assigned to the LT waitlist
* English-speaking
* No contraindication to moderate intensity physical activities
* Physician clearance for participation in moderate intensity physical activities
* No history of dementia or organic brain syndrome

Caregivers:

* Adult (age≥ 19 years)
* English-speaking
* Provide direct care to LT candidates

Exclusion Criteria:

* Inability to communicate verbally in English
* Documentation of cognitive deficits

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult, all gender, and all race patients with end-stage liver disease (ESLD) who have been assigned to the liver transplant (LT) waitlist. Nationally, the median age of LT candidates is 57 (48, 63) during 2014 to 2018. UAB Liver Transplant Center technically does not limit patients over 75 years old for LT (i.e., age alone is not an absolute contraindication), but typically as patients age they have less physiologic reserve to tolerate transplant so they must have a better pre-transplant functional status than a younger patient in order to have a good outcome post-transplant. Participants will be identified and recruited from the UAB Liver Transplant Center using a purposive maximum variation sampling approach in terms of age, gender, race, and severity of ESLD.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Liver frailty index (LFI) score | From baseline through 3 months
  Change from baseline in liver frailty index score at 3 months; the higher LFI scores indicate a higher degree of frailty. LFI<3.2: robust, LFI=3.2-4.4: prefrail, LFI>=4.5: Frail.
Caregiver burden measured using Zarit Burden Interview short form (ZBI-12) | From baseline through 3 months
  Change from baseline in the total ZBI-12 scores at 3 months. The total ZBI-12 score is the summation of 12 items, ranging from 0 to 48; the higher scores indicate higher burden (0-10:no to mild burden; 10-20: mild to moderate burden), and >20: high burden.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Qu, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
The nominal group technique meeting data will be shared in an aggregate level by group. The card-sorting data and rating data will be shared in an aggregate level by participant type (patient vs caregiver).